CLINICAL TRIAL: NCT01168817
Title: A Prospective, Randomized, Double-blind, Double-dummy, Placebo- and Active Controlled, Multicenter Study Assessing the Efficacy and Safety of the Combination BAY60-4552 / Vardenafil Compared to Vardenafil (20 mg) for the Treatment of Erectile Dysfunction Not Sufficiently Responsive to Standard Therapy With PDE5 (Phosphodiesterase 5) Inhibitors
Brief Title: Clinical Proof-of-concept Study for the Combination BAY60-4552 / Vardenafil for the Treatment of Erectile Dysfunction Not Sufficiently Responsive to Standard Therapy With PDE5 Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14694; 2010-020122-18 (EudraCT Number)
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Erectile Dysfunction
Keywords: Combination Drug Therapy; Phosphodiesterase inhibitors
MeSH Terms: conditions — Erectile Dysfunction | interventions — BAY 60-4552; Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: BAY60-4552 plus Vardenafil
- Arm 2 (Active Comparator)
  Interventions: Drug: Vardenafil
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY60-4552 plus Vardenafil — Treatment with 3 tablets once daily for 4 weeks (Vardenafil 10 mg plus BAY60-4552 1.0 mg)
  Arms: Arm 1
Drug: Vardenafil — Treatment with 3 tablets once daily for 4 weeks (Vardenafil 20 mg)
  Arms: Arm 2
Drug: Placebo — Treatment with 3 tablets once daily for 4 weeks (Placebo)
  Arms: Arm 3

SUMMARY:
This study examines the efficacy and safety of the combination treatment BAY60-4552 plus vardenafil in patients with erectile dysfunction, who do not sufficiently respond to therapy with PDE5 (Phosphodiesterase 5) inhibitors.

Patients meeting the entry criteria, will receive vardenafil alone in the first four weeks of the study to assess the effect of PDE5 inhibitor therapy given alone.

Patients with an insufficient therapeutic response to vardenafil alone will enter the next part of the study, and will be randomly assigned to one of 3 treatments. There is a 1 in 3 chance of receiving either the combination BAY60-4552 plus vardenafil, or vardenafil alone, or placebo. Neither patient nor the treating physician will know which treatment is given (double-blinded design).This part of the study will last four weeks Patients will have to go to the clinic/hospital for 7 visits during the 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Open-label run-in phase (first four weeks):

  * Written informed consent signed before any study-specific procedure
  * History of ED (Erectile Dysfunction) for at least 6 months prior to screening, defined as "the inability to achieve and maintain an erection of the penis sufficient to complete satisfactory sexual intercourse"; the diagnosis of ED has to be confirmed by a physician
  * Stable, heterosexual relationship for at least 6 months prior to screening
  * Aged 18 to 64 years (inclusive) at the first screening examination
  * History of previous use of at least 1 marketed PDE5 (Phosphodiesterase 5) inhibitor and insufficient therapeutic efficacy despite use of the highest approved dose
* Double-blind treatment phase (last four weeks):

  * At least 4 attempts at sexual intercourse on 4 separate days during the open-label run-in phase with use of 20 mg vardenafil approximately 1 hour before attempting intercourse
  * IIEF EF (International Index of Erectile Function - Erectile Function subscale) score <17
  * At least 50% of attempts at sexual intercourse during the open-label run-in phase were unsuccessful

Exclusion Criteria:

* Contraindication to use of vardenafil
* History of prostatectomy due to prostate cancer, including nerve-sparing techniques.
* Concomitant use of adrenergic blockers
* History of spinal cord injury
* Resting hypotension, i.e. SBP (Systolic Blood Pressure) <100 mmHg at rest
* Moderate / severe hypertension, i.e. SBP >170 mmHg or DBP >110 mmHg at rest
* Symptomatic orthostatic hypotension with a decrease in SBP >20 mmHg or in DBP (Diastolic Blood Pressure) >10 mmHg subsequent to change from the supine to standing position

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Severity of erectile dysfunction assessed by the IIEF-EF (International Index of Erectile Function - Erectile Function subscale) | Week 4

SECONDARY OUTCOMES:
Success rate assessed by subject diary question: 'Maintenance' (Did your erection last long enough to have sexual intercourse?) | Week 4
Success rate assessed by subject diary question: Penetration' (Were you able to insert your penis into your partner's vagina?) | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (33):
- Finland (3):
  - Oulu
  - Tampere
  - Turku
- France (6):
  - Chambéry
  - Garches
  - Lille
  - Lyon
  - Nice
  - Nîmes
- Germany (7):
  - Weiden, Bavaria
  - Hamburg, Hamburg
  - Marburg, Hesse
  - Osnabrück, Lower Saxony
  - Mülheim, North Rhine-Westphalia
  - Koblenz, Rhineland-Palatinate
  - Leipzig, Saxony
- Italy (4):
  - Florence
  - Milan
  - Napoli
  - Roma
- Netherlands (3):
  - Groningen, Provincie Groningen
  - Leiden
  - The Hague
- Spain (4):
  - Barcelona, Barcelona
  - Aravaca, Madrid
  - Majadahonda, Madrid
  - Málaga, Málaga
- Sweden (6):
  - Eskilstuna
  - Gothenburg
  - Halmstad
  - Jönköping
  - Linköping
  - Stockholm

REFERENCES:
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu